CLINICAL TRIAL: NCT06021496
Title: The Effect of Two Different Methods of Health Education on Women's HPV Knowledge, Cervical Cancer Health Belief and Screening
Brief Title: The Effect of Face-to-face and Online Health Education on Women's Cervical Cancer Knowledge, Health Beliefs and Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, Asisstant Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CERVİCAL CANCER
Record Dates: First submitted 2023-08-18; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Early Detection of Cancer
Keywords: Cervical Cancer; Cervical Cancer Screening; Health Education; Online Education; Home Visit
MeSH Terms: conditions — Uterine Cervical Neoplasms; Health Education

STUDY DESIGN:
Intervention Model Description: randomised control trial
Who Masked: Participant
Masking Description: single blind study, participants do not know their group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Participants in the control group continued to receive standard cervical cancer screening service of the Ministry of Health. No further intervention was made.
- Face-to-face training group (Experimental): In addition to the standard cervical screening service of the Ministry of Health, face-to-face health education through home visits and a reminder by phone call were made once.
  brochure given
  Interventions: Behavioral: face to face health education
- Online training group (Experimental): In addition to the standard cervical screening service of the Ministry of Health, online health education via video call and a reminder with a phone call once. A digital brochure was given.
  Interventions: Behavioral: online health education

INTERVENTIONS:
Behavioral: face to face health education — Face-to-face health education with home visit
  Arms: Face-to-face training group
Behavioral: online health education — online health education with video call
  Arms: Online training group

SUMMARY:
Aim: The aim of this study is to determine the effect of health education given by two different methods on women's knowledge about HPV, cervical cancer health belief and screening test.

Materials and Methods: The study was conducted in a parallel groups design as a single-blind randomized controlled trial. The sample consisted of 126 healthy participants, 42 in each volunteer group, who were registered at the Martyr Zafer Çalışkan Family Health Center in Ankara between January and July 2023, and met the inclusion criteria. HPV Knowledge scale, Cervical Cancer and pap Smear Test Health Belief Model Scale and VAS for self-assessment were used in the study. In the study, while the control group received standard care, the face-to-face education group was given health education and brochures through home visits and a reminder interview over the phone; On the other hand, the online training group was given health education and a digital brochure via video call and a reminder meeting was held once. One-way analysis of variance and Kruskal Wallis test were used to compare the data of the three groups after a two-month follow-up, Tukey and Dunn test for multiple comparisons, and Wilcoxon test for in-group comparisons before and after. In addition, two-way analysis of variance and Robust ANOVA were used in group and time comparisons.

DETAILED DESCRIPTION:
In this randomized controlled trial, participants were assigned to three groups by the block randomization method and the study was conducted in a single-blind parallel groups design. It was carried out at Martyr Zafer Çalışkan Family Health Center between January 2023 and July 2023. The eligibility of female participants between the ages of 30-65 to participate in the study was evaluated by the researcher. The sample size was calculated based on the rate of cervical cancer screening test in Kurt and Akyüz's study. G Power 3.1.9.2 package program was used in the calculation. Taking into account possible data loss, it was decided to add 30% backup participants. In this context, the sample of the study was calculated as 126 participants, 42 in each group. The patients who volunteered to participate in the study were examined whether they met the inclusion criteria other than the level of drug compliance. Written informed consent was obtained from the participants who met the inclusion criteria and a questionnaire form was applied. Participants were assigned to groups using the block randomization method. No intervention was made in the control group. At the end of the following first week, face-to-face and online training was provided with the participants in the online training group, one-to-one home visits, face-to-face training and video calls. Four weeks later, a brief reminder was made by phone call. At the end of eight weeks, a second questionnaire was applied to all groups.

ELIGIBILITY:
The criteria for inclusion in this study are;

1. Volunteering to participate in the study,
2. To be between the ages of 30-65,
3. Being a woman
4. Being married/having an active sexual life,
5. Having the technical equipment to make video calls,
6. To be literate in Turkish,
7. Not having had an HPV DNA / Pap Smear test in the last 5 years. -

Exclusion Criteria:

The criteria for not being included in this study are;

1. Being pregnant or in the postpartum trimester,
2. Having a family history of cervical cancer,
3. Having had a hysterectomy operation,
4. To have received any previous training on cervical cancer,
5. Having a vaginal infection,
6. To be vaccinated against HPV (3 doses). -

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — intervention for cervical cancer
Enrollment: 126 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
HPV Knowledge Scale | 60 days
  HPV Knowledge Scale consists of 4 sub-dimensions and 33 items. Participants score between 0-33.

SECONDARY OUTCOMES:
Cervical Cancer and Pap Smear Test Health Belief Model Scale | 60 days
  Although the scale is graded in a 5-point Likert type, it consists of a total of 35 items. The higher the scores obtained from the scale, the higher the sensitivity, caring and motivation; It means that benefits are perceived high for the perception of benefit, and obstacles are perceived high for the perception of obstacles.

CONTACTS AND LOCATIONS:
Overall Officials: merve gökmen, Principal Investigator — Ministry of Health
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No